CLINICAL TRIAL: NCT07252310
Title: Pilot Study of Acceptability and Feasibility of StudyU for N-of-1 Trials
Brief Title: Pilot Study of StudyU for N-of-1 Trials in HFrEF Patients (N-of-1 App)
Acronym: N-of-1 App
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-08029225
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: HFrEF - Heart Failure With Reduced Ejection Fraction; Heart Failure; Heart Failure, Systolic; Heart Diseases
Keywords: HFrEF; App; N-of-1; GDMT; StudyU; Beta Blocker
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Diseases; Alzheimer Disease | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- GDMT (Beta Blockers) (Experimental): This study consists of a single arm. Subjects will complete study activities remotely. Following enrollment, daily assessments will be conducted using the StudyU mobile application. Additional assessments will occur at the end of each study period, completed by phone, WCM Zoom, or via email, depending on subject preference. The study involves testing multiple doses of each subject's guideline-directed medical therapy (GDMT), specifically beta-blockers. Doses will include the subject's current home dose (as prescribed by their treating physician prior to enrollment), as well as one or more increased -and, if needed, decreased-doses that are near or at the guideline-directed maximum. All dosing decisions will be made collaboratively by the PI, the subject's clinician, and the participant, taking into account titration guidelines, physician guidance, and subject symptoms and preferences. Each subject will complete a minimum of two periods. The number of periods is adaptive.
  Interventions: Drug: beta blockers; Device: StudyU Application

INTERVENTIONS:
Drug: beta blockers — Subjects will remain on their current home dose of beta blocker (as prescribed by their treating physician prior to enrollment) during Period 1. In Period 2, the dose will be increased -either doubled or by 50%-to support progression toward the guideline-directed medical therapy (GDMT) target. may choose to continue on the tested dose and conclude the study, or request additional information before selecting their preferred dose. If both the participant and the study clinician agree that further evaluation is needed, a third period will be initiated. In this period, the dose may again be increased-by 50% or doubled relative to the Period 2 dose-if tolerated and agreed upon by the participant. If the new dose is well-tolerated and the participant agrees to continue with dose escalation after reviewing their data, the dose will be increased again-either doubled or increased by 50%-for the next period (Period 3). The study team will continue to collect data.
Device: StudyU Application — StudyU is a novel mobile app developed for the design of and conduct of N-of-1 trials. StudyU consists of the StudyU Designer, a web platform and mobile app, accessible through the website https://designer.studyu.health; the StudyU App for smartphones, which can be downloaded from Apple and Google app stores, and the secure backend where data is stored. All components of StudyU were developed by Dr. Stefan Konigorski and his colleagues at Hasso-Plattner Institute (HPI) for Digital Engineering at the University of Potsdam. The StudyU platform allows investigators to easily operationalize their study processes in the StudyU designer. In the StudyU designer, investigators indicate at which frequency subjects will complete assessments. For this pilot trial, a WCM-specific instance of StudyU will be developed and hosted on the secure WCM server. Only the WCM study team will have access to the subject data from the StudyU App.

SUMMARY:
This study will look at whether using a phone app called StudyU can help people with Heart Failure with Reduced Ejection Fraction (HFrEF) reach their recommended dose on their beta blocker.

DETAILED DESCRIPTION:
The overarching goal of this study is to determine feasibility of the StudyU app in N-of-1 trials. The study intervention is N-of-1 trials, facilitated by a mobile-based application, StudyU. The study team will utilize a single-arm sequential design N-of-1 study in which subjects who are not yet at the GDMT for beta blockers will test multiple doses of GDMT to understand the maximally tolerated dose using an N-of-1 trial format. This is similar to an approach used in a previous study, Pilot Deprescribing N-of-1 Trials for beta blockers in HFpEF (NCT04757584) but will test the addition of a mobile-based app to collect vital signs, monitor side effects, and monitor patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 65 years old
2. A history of HFrEF per electronic medical record review/clinician impression that is defined as an EF <50% that is shown from any imaging modality
3. Taking less than the maximal dose of beta blocker per physician recommendation at time of enrollment
4. Access to a smartphone or device that can perform many of the same functions as a computer, typically having a touchscreen interface, internet access, and an operating system capable of running downloaded applications

Exclusion Criteria:

1. Clinical instability (this N-of-trial is appropriate for stable conditions only)

   1. Decompensated HF
   2. Hospitalized in the past 30 days
   3. Medication changes or procedures in prior 14 days (to prevent confounding from other interventions) at PI discretion
2. Do not have access to a smartphone or tablet
3. Estimated life expectancy <6 months
4. Moderate-severe dementia or psychiatric disorder precluding informed consent
5. Language barrier that will preclude informed consent and ability to comprehend study procedures
6. History of noncompliance or inability to complete study procedures
7. Enrollment in a clinical trial not approved for co-enrollment
8. Any condition that, in Principal Investigator or treating physician's opinion, makes the patient unsuitable for study participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure Score | End of intervention visit, assessed between Week 6 (minimum) and Week 18 (maximum).
  The Feasibility of Intervention (FIM) measure is a survey that evaluates an intervention's practicality. Questions are ranked on 1- to 5-point Likert scales, with higher scores indicating higher feasibility and lower indicating less feasibility. Total scores range from 4 to 20. A score of 4 indicates low feasibility and a score of 20 indicates strong feasibility.
Intervention Appropriateness Measure Score | End of intervention visit, assessed between Week 6 (minimum) and Week 18 (maximum).
  The Intervention Appropriateness Measure (IAM) is a survey that evaluates an intervention's suitability and compatibility. Questions are ranked on 1- to 5-point Likert scales, with higher scores indicating higher appropriateness and lower indicating less appropriateness. Total scores range from 4 to 20. A score of 4 indicates low appropriateness and a score of 20 indicates strong appropriateness.
Acceptability of Intervention Measure Score | End of intervention visit, assessed between Week 6 (minimum) and Week 18 (maximum).
  Acceptability of Intervention Measure (AIM) is a survey that evaluates how agreeable an intervention is to participants. Questions are ranked on 1- to 5-point Likert scales, with higher scores indicating higher acceptability and lower indicating less acceptability. Total scores range from 4 to 20. A score of 4 indicates low acceptability and a score of 20 indicates strong acceptability.

SECONDARY OUTCOMES:
Change in KCCQ-12 Score | Baseline, assessed on Day 1. End of Period visit, assessed between Week 3 (minimum) and Week 18 (maximum). End of intervention visit, assessed between Week 6 (minimum) and Week 18 (maximum).
  The Kansas City Cardiomyopathy Questionnaire-12 (KCCQ) is a heart failure-specific health status survey. Questions are ranked on 5- to 7-point Likert scales, with higher scores indicating better health status and lower indicating worse health status. Total scores range from 0 to 100. A score of 0 indicates the worst health statues and a score of 100 indicates the best health status score. The change in score is comparing the baseline dose with the changed dose in subsequent periods. End of Period visits can convert to end of intervention if participants choose that dose.
Change in PROMIS-29 Score | Baseline, assessed on Day 1. End of Period visit, assessed between Week 3 (minimum) and Week 18 (maximum). End of intervention visit, assessed between Week 6 (minimum) and Week 18 (maximum).
  Patient-Reported Outcome Measurement Information System-29 (PROMIS) is a health-related quality of life survey, with questions from 7 domains: depression, anxiety, physical function, pain interference, pain intensity, sleep disturbance, and ability to engage in social roles and activities. Questions are ranked on a 5-point Likert scale, with higher scores at times indicating better quality of life, and lower scores indicating poorer quality of life. Scores are reported for each domain. Total scores range for each domain except pain intensity is from 0 to 100. A score of 0 indicates no symptoms, whereas a 100 indicates extremely severe symptoms for each domain. For the pain intensity domain, there is a pain rating scale from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. The change in score is comparing the baseline dose with the changed dose in subsequent periods. End of Period visits can convert to end of intervention if participants choose that dose.
Change in PROMIS CF-SF 6a Score | Baseline, assessed on Day 1. End of Period visit, assessed between Week 3 (minimum) and Week 18 (maximum). End of intervention visit, assessed between Week 6 (minimum) and Week 18 (maximum).
  Patient-Reported Outcome Measurement Information System Cognitive Function - Short Form 6a (PROMIS CF-SF) Score is a health-related quality of life survey that focuses on the cognitive function domain. Questions are ranked on a 5-point Likert scale, with higher scores at times indicating higher cognitive function, lower scores indicate lower cognitive function. Total scores range from 0 to 100. A score of 0 indicates worst possible cognitive function, whereas a 100 indicates best possible cognitive function. The change in score is comparing the baseline dose with the changed dose in subsequent periods. End of Period visits can convert to end of intervention if participants choose that dose.
Change in PROMIS Sexual Function Score | Baseline, assessed on Day 1. End of Period visit, assessed between Week 3 (minimum) and Week 18 (maximum). End of intervention visit, assessed between Week 6 (minimum) and Week 18 (maximum).
  Patient-Reported Outcome Measurement Information System (PROMIS) Sexual Function Score is a health-related quality of life survey that focuses on the sexual function domain. Questions are ranked on a 5-point Likert scale, with higher scores at times indicating higher sexual function, lower scores indicate lower sexual function. Total scores range from 0 to 100. A score of 0 indicates no sexual interest/function/satisfaction whereas a 100 indicates high sexual interest/function/satisfaction. The change in score is comparing the baseline dose with the changed dose in subsequent periods. End of Period visits can convert to end of intervention if participants choose that dose.

CONTACTS AND LOCATIONS:
Overall Officials: Parag Goyal, MD, MSc, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goyal P, Safford MM, Hilmer SN, Steinman MA, Matlock DD, Maurer MS, Lachs MS, Kronish IM. N-of-1 trials to facilitate evidence-based deprescribing: Rationale and case study. Br J Clin Pharmacol. 2022 Oct;88(10):4460-4473. doi: 10.1111/bcp.15442. Epub 2022 Jul 13. PMID 35705532
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Verhestraeten C, Heggermont WA, Maris M. Clinical inertia in the treatment of heart failure: a major issue to tackle. Heart Fail Rev. 2021 Nov;26(6):1359-1370. doi: 10.1007/s10741-020-09979-z. PMID 32474794
- [Background] Rao VN, Greene SJ. Breaking Clinical Inertia in Heart Failure Management. Jt Comm J Qual Patient Saf. 2022 Jan;48(1):3-4. doi: 10.1016/j.jcjq.2021.11.002. Epub 2021 Nov 11. No abstract available. PMID 34840128